CLINICAL TRIAL: NCT01907334
Title: Dose-response of Salmeterol Delivered by Advair Diskus in Children: Bioassay by Methacholine Challenge Using Oscillometry as the Endpoint
Brief Title: Dose-Response of Salmeterol in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 38-2013
Record Dates: First submitted 2013-06-28; First posted 2013-07-24 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Asthma
Keywords: oscillometry; asthma; methacholine
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Methacholine Chloride; Albuterol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advair Diskus100/50 µg and Advair Diskus 100/50 µg (Active Comparator): The Advair Diskus 100/50 µg and Advair Diskus 100/50 µg will be administered in a blinded fashion. One hour after receiving the dose of Advair a methacholine challenge will be performed to determine the PC40R5. After the PC40R5 has been reached or a negative result after the highest methacholine concentration, 64 mg/mL, subjects will inhale albuterol through a valved holding chamber to reverse bronchoconstriction and their lung function will be monitored until it has returned to within 20% of that day's baseline R5.
  Interventions: Drug: Advair Diskus100/50 µg; Drug: Methacholine Chloride; Drug: Albuterol
- Advair Diskus 100/50 µg and Flovent Diskus 100 µg (Active Comparator): The Advair Diskus 100/50 µg and Flovent Diskus 100 µg will be administered in a blinded fashion. One hour after receiving the dose of Advair and Flovent a methacholine challenge will be performed to determine the PC40R5. After the PC40R5 has been reached or a negative result after the highest methacholine concentration, 64 mg/mL, subjects will inhale albuterol through a valved holding chamber to reverse bronchoconstriction and their lung function will be monitored until it has returned to within 20% of that day's baseline R5.
  Interventions: Drug: Advair Diskus100/50 µg; Drug: Flovent Diskus 100 µg; Drug: Methacholine Chloride; Drug: Albuterol

INTERVENTIONS:
Drug: Advair Diskus100/50 µg — Advair Diskus 100/50 µg
  Other Names: fluticasone; salmeterol
Drug: Flovent Diskus 100 µg — Flovent Diskus 100 µg
  Other Names: fluticasone
  Arms: Advair Diskus 100/50 µg and Flovent Diskus 100 µg
Drug: Methacholine Chloride — Methacholine Chloride in quadrupling concentrations from 0.25 to 64 mg/mL will be given based upon subject's baseline response.
Drug: Albuterol — Albuterol will be administered at the end of each methacholine challenge.

SUMMARY:
To examine whether a breathing test (methacholine challenge using impulse oscillometry) can be used to tell the difference between two different doses of an inhaled drug, salmeterol, delivered by Advair in children with asthma

DETAILED DESCRIPTION:
During the study the subject will have to attend 4 study visits: 2 screening visits and 2 treatment visits.

Before each study visit, the subject has to stop using certain asthma medications.

At Screening Visit 1a, the parent/guardian will read and sign the informed consent form to allow the subject to take part in this study. The subject, if appropriate, will be asked to sign the last page to indicate his/her assent to be in the study.

The study coordinator will conduct an interview to find out about the subject's medical history, diseases other than asthma, previous medication and any medication that the subject will take during his/her participation in this study. Vital signs, i.e. blood pressure, heart rate, and respiration, and height and weight will be measured, and an electrocardiogram (ECG) which is a test to measure the electrical activity of the subject's heart, will be performed. The subject will be examined by a Pediatric Pulmonary physician and will be taught the proper way to use a Diskus® inhaler. The subject has to be able to show that he/she can do this correctly.

At Screening Visit 1b, if all of the tests are in the appropriate range the subject will take 2 puffs of Flovent from a Diskus®. One hour later, the subject will perform a breathing test called impulse oscillometry. Essentially, a sound is sent down into the lungs and a computer converts the return sound into a number. Then the subject will begin a breathing test with methacholine, a drug that makes the airways smaller. He/she will begin by inhaling a low dose in a nebulizer and then performing oscillometry. After a 5 minute interval he/she will breathe in increasing doses, up to 6 times or until his/her breathing test increases by 40%. Albuterol will be administered immediately after the end of the challenge and the subject will be monitored until his/her breathing returns to within 20% of where it was before the challenge.

If the methacholine test results are within the appropriate range the subject will be eligible for the treatment phase and will be scheduled for Visit No. 2.

At each treatment visit, the subject will take 2 puffs of study drug from two Diskus® inhalers, either 1 puff of Flovent and 1 puff of Advair, or 1 puff of Advair from two different inhalers. This is done in a blinded manner so the study coordinator does not know which treatment is used each time. There will be a 1 hour wait time after the medication is administered before the methacholine challenge is started. Albuterol will be administered immediately after the end of the challenge and the subject will be monitored until his/her breathing returns to within 20% of where it was before the challenge.

ELIGIBILITY:
Inclusion Criteria:

* parent/legal guardian and subject must be able to speak and understand English and patient must be willing and able to give assent to take part in the study
* diagnosed with asthma for at least 6 months
* able to demonstrate inhalation technique with study device
* if taking inhaled corticosteroids, dose must be stable for 2 weeks
* no significant concomitant medical conditions or abnormal physical findings on screening except for those consistent with asthma and allergic rhinitis
* airway responsiveness to methacholine with a baseline provocational dose causing an increase of at least 40% in R5 (PC40R5) at no more than 8 mg/mL

Exclusion Criteria:

* female who has started menstruating
* past or present history of any allergic reaction to any of the medications or formulations administered in this study
* prior treatment with systemic corticosteroids in last 30 days or more than 4 courses in previous 12 months
* use of short-acting beta-agonist more than two times per week in the previous month
* use of long-acting beta-agonist in the 3 weeks before the first methacholine challenge or during the study
* change in dosage of inhaled corticosteroids in previous 30 days, nasal steroids in previous 15 days and montelukast in last 7 days
* history of life-threatening asthma, including loss of consciousness, intubation and/or admission to ICU
* hospitalization for acute asthma within past year
* inability to withhold the following medications before methacholine challenges:
* short-acting beta-agonists at least 6 hours
* regular long-acting beta-agonists at least 3 weeks
* inhaled corticosteroid at least 2 hours
* montelukast at least 24 hours
* aspirin and non-steroid anti-inflammatory drugs at least 48 hours
* caffeine at least 4 hours

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hendeles, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Asthma Research Lab, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Advair and Advair Diskuses, Then Advair and Flovent Diskuses: On treatment day one, Advair 100/50 mcg and Advair 100/50 mcg were administered in a blinded fashion. One hour after receiving the dose a methacholine challenge was performed to determine PC40R5. After PC40R5 was reached or a negative result after the highest methacholine concentration, 64 mg/mL, subjects inhaled albuterol through a valved holding chamber to reverse bronchoconstriction and their lung function was monitored until it returned to within 20% of that day's baseline R5.
  On treatment day two, Advair 100/50 mcg and Flovent 100 mcg were administered in a blinded fashion. One hour after receiving the dose a methacholine challenge was performed to determine PC40R5. After PC40R5 was reached or a negative result after the highest methacholine concentration, 64 mg/mL, subjects inhaled albuterol through a valved holding chamber to reverse bronchoconstriction and their lung function was monitored until it returned to within 20% of that day's baseline R5.
- Advair and Flovent Diskuses, Then Advair and Advair Diskuses: On treatment day one, Advair 100/50 mcg and Flovent 100 mcg were administered in a blinded fashion. One hour after receiving the dose a methacholine challenge was performed to determine PC40R5. After PC40R5 was reached or a negative result after the highest methacholine concentration, 64 mg/mL, subjects inhaled albuterol through a valved holding chamber to reverse bronchoconstriction and their lung function was monitored until it returned to within 20% of that day's baseline R5.
  On treatment day two, Advair 100/50 mcg and Advair 100/50 mcg were administered in a blinded fashion. One hour after receiving the dose a methacholine challenge was performed to determine PC40R5. After PC40R5 was reached or a negative result after the highest methacholine concentration, 64 mg/mL, subjects inhaled albuterol through a valved holding chamber to reverse bronchoconstriction and their lung function was monitored until it returned to within 20% of that day's baseline R5.
Period: Overall Study
Arm/Group | Advair and Advair Diskuses, Then Advair and Flovent Diskuses | Advair and Flovent Diskuses, Then Advair and Advair Diskuses
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were analyzed according to protocol.
Groups:
- All Participants: Participants were randomized to either Advair 100/50 mcg and Advair 100/50 mcg, then Advair 100/50 mcg and Flovent 100 mcg OR Advair 100/50 mcg and Flovent 100 mcg, then Advair 100/50 mcg and Advair 100/50 mcg.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Airway Resistance Increase
Description: concentration of methacholine required to increase total airway resistance by 40% (PC40R5)
Time Frame: 1 to 7 days
Population: The analysis was performed on all 10 participants.
Measure: Geometric Mean (95% Confidence Interval); unit: ln(mg/mL)
Groups:
- Increase in Airway Resistance After Methacholine: Participants were randomized to either Advair 100/50 mcg and Advair 100/50 mcg, then Advair 100/50 mcg and Flovent 100 mcg OR Advair 100/50 mcg and Flovent 100 mcg, then Advair 100/50 mcg and Advair 100/50 mcg. On each study day after treatment, methacholine challenge was performed to determine provocational concentration of methacholine which caused a 40% increase in resistance at 5 Hz (PC40R5).
Arm/Group | Increase in Airway Resistance After Methacholine
Number analyzed (Participants) | 10
ln(mg/mL)
  Advair and Advair Diskuses | 47 [25.18 to 87.78]
  Advair and Flovent Diskuses | 22.9 [8.48 to 61.61]

ADVERSE EVENTS:
Arm/Group | Advair and Advair Diskuses, Then Advair and Flovent Diskuses | Advair and Flovent Diskuses, Then Advair and Advair Diskuses
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No